CLINICAL TRIAL: NCT04313413
Title: Effectiveness of Yoga@Work Program for Reducing Musculoskeletal Pain in Neck and Shoulder: Evaluation Study
Brief Title: Yoga@Work for Reducing Musculoskeletal Pain in Neck and Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Brunel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU03
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Neck Pain; Shoulder Pain; Musculoskeletal Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Musculoskeletal Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga@Work (Experimental): Yoga sessions specifically designed for office workers were provided in work settings. participants were given handouts and encouraged to practice in their own time and space during work days.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Yoga sessions includes sukshma vyayama (strengthening yoga expertise), stretching and relaxing postures (asana) on chair or standing, breathing and meditation practices.

SUMMARY:
Work-related musculoskeletal disorders (MSDs) are disorders of muscles, tendons, joints and nerves which can affect all body parts, although the neck, upper limb and back are the most common areas.

The peer-reviewed literature about workplace prevention describes a variety of interventions that have been implemented and evaluated.but only few studies show sustainable positive effects on symptom outcomes.

Yoga@Work program was developed to self manage pain around neck and shoulder areas among office workers.

ELIGIBILITY:
Inclusion Criteria:

* Office workers
* Willing to participate and give consent
* non specific neck and shoulder pain

Exclusion Criteria:

* neck injury
* Trauma
* Cancer related pain
* psychiatric disorder/ medication
* Pregnancy

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Neck and Shoulder pain | From baseline to 4-week post intervention
  self reported neck and shoulder pain using visual analogue scale on 0 to 10 scale, where 0 is no pain and 10 is worst pain.

SECONDARY OUTCOMES:
Global Outcome | from baseline to 5 week post intervention
  Patient Global Received Rating of Improvement or Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK; Monomita Nandy, Study Chair — Brunel University
Locations (1):
- Yog Kulam, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided